CLINICAL TRIAL: NCT05505773
Title: Prospective Clinical Study to Evaluate the Metabolism Using the Breezing Device in the Preoperative and Postoperative Periods of Gastric Bypass in Patients With Type II Diabetes.
Brief Title: Systemic Metabolic Rate of Diabetic Patients Before and After Bariatric Gastric Bypass Using the Breezing® Device.
Status: Completed | Type: Observational
Sponsor: Kaiser Clinic and Hospital (Other)
Responsible Party: Principal Investigator, Luiz Gustavo de Quadros, MD, Prospective Clinical Study to Evaluate the Metabolism Using the Breezing Device in the Preoperative and Postoperative Periods of Gastric Bypass in Patients With Type II Diabetes., Kaiser Clinic and Hospital
Other Study IDs: Breezing
Record Dates: First submitted 2022-08-16; First posted 2022-08-18 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Obesity; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity; Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To evaluate the systemic metabolic rate of diabetic patients before and after bariatric gastric bypass surgery using the Breezing® device.

DETAILED DESCRIPTION:
Objective of the research:

Primary To evaluate the systemic metabolic rate of diabetic patients before and after bariatric gastric bypass surgery using the Breezing® device.

Secondary

* To measure the indirect metabolic rate by quantifying O2 gas consumption (g) and CO2 gas release (g);
* To analyze the 'population impact', that is, to measure using statistical tools how many cases of metabolic maladjustment could be prevented if the diabetes risk factor were to be eliminated;
* To correlate, by means of a regression test, if there is any dependence between the metabolic rate and the diabetes risk factor;
* To validate the accuracy of the Breezing® device.

Evaluation of the risks and benefits Risks As the patient only needs to blow on the Breezing® device using a small straw (blower), the direct risks are minimal, perhaps contamination due to failure to exchange the blower. Thus, the risks are indirect and are more associated to the malfunctioning of the device.

Benefits The advantage is that the procedure is simple and can provide results with important information about the metabolic rate even just using the iPhone or iPad of patients as a strategy to monitor metabolic control.

ELIGIBILITY:
Inclusion Criteria: over 18 years -

Exclusion Criteria: obesity

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: obesity
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2019-01-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the systemic metabolic rate of diabetic patients before and after bariatric gastric bypass surgery using the Breezing® device. | 2 years
  metabolic rate of diabetic patients before and after bariatric gastric bypass surgery using the Breezing® device.

CONTACTS AND LOCATIONS:
Overall Officials: Luiz Gustavo de Quadros, MD, Principal Investigator — Kaiser Clinica and Day Hospital